CLINICAL TRIAL: NCT00098670
Title: A Phase II Study of Fludarabine + Rituximab Induction Followed by Alemtuzumab (Campath-1H, NSC #715969, IND #10864) Administered Subcutaneously as Consolidation in Untreated Patients With B-Cell Chronic Lymphocytic Leukemia
Brief Title: Fludarabine, Rituximab, and Alemtuzumab in Treating Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02812; NCI-2012-02812 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000398139; CALGB-10101 (Other: Cancer and Leukemia Group B); CALGB-10101 (Other: CTEP); P30CA014236 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Results first posted 2012-12-03 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2012-12

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Stage I Chronic Lymphocytic Leukemia; Stage II Chronic Lymphocytic Leukemia; Stage III Chronic Lymphocytic Leukemia; Stage IV Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab; Rituximab; fludarabine phosphate

ARMS (1):
- Treatment (alemtuzumab, rituximab, fludarabine phosphate) (Experimental): Patients receive induction therapy comprising rituximab IV over 4 hours on days 1, 3, and 5 of course 1 and day 1 of all subsequent courses and fludarabine IV over 30 minutes on days 1-5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression.
  Approximately 4 months after completion of induction therapy, patients achieving a partial response, nodular partial response, or stable disease receive consolidation therapy comprising alemtuzumab subcutaneously on days 1-3. Treatment repeats weekly for up to 6 courses in the absence of disease progression.
  Interventions: Biological: alemtuzumab; Biological: rituximab; Drug: fludarabine phosphate

INTERVENTIONS:
Biological: alemtuzumab — Given SC
  Other Names: anti-CD52 monoclonal antibody; Campath-1H; MoAb CD52; Monoclonal Antibody Campath-1H; Monoclonal Antibody CD52
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara

SUMMARY:
This phase II trial is studying how well giving fludarabine together with rituximab followed by alemtuzumab works in treating patients with chronic lymphocytic leukemia. Monoclonal antibodies, such as rituximab and alemtuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others can find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as fludarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving fludarabine together with rituximab followed by alemtuzumab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the rate of complete response and toxicity of concurrent treatment with fludarabine and rituximab followed by consolidative alemtuzumab in patients with previously untreated, but symptomatic, CLL.

II. To determine if alemtuzumab improves the CR rate with acceptable toxicity when administered as consolidation therapy following induction therapy with fludarabine and rituximab.

III. To estimate the progression-free and overall survival of high risk (VH gene unmutated and those with p53 dysfunction) and low-risk (others) patients following therapy with fludarabine and rituximab induction and consolidative alemtuzumab.

IV. To determine the frequency of molecular (PCR) remission following fludarabine and rituximab induction therapy and alemtuzumab consolidation therapy and if this serves as a surrogate marker for prolonged progression-free and overall survival.

SECONDARY OBJECTIVES:

I. To determine the effect of concurrent treatment with fludarabine and rituximab followed by consolidative alemtuzumab on recovery of T-cells, NK cells, and serum immunoglobulin levels.

II. To determine clinical and molecular features that predict for poor response to fludarabine and rituximab induction and subsequent alemtuzumab consolidation therapy.

III. To assess preliminarily the molecular features of CLL at relapse in patients responding to chemoimmunotherapy for CLL.

IV. To determine the frequency of patients who remain at high risk for progression of CLL despite this therapy and who are thus eligible for nonmyeloablative stem cell transplantation studies such as CALGB 109901.

V. To perform limited rituximab pharmacokinetics to determine the ideal schedule of administration for a subsequent rituximab maintenance treatment approach following induction therapy with fludarabine and rituximab.

OUTLINE:

Patients receive induction therapy comprising rituximab IV over 4 hours on days 1, 3, and 5 of course 1 and day 1 of all subsequent courses and fludarabine IV over 30 minutes on days 1-5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression.

Approximately 4 months after completion of induction therapy, patients achieving a partial response, nodular partial response, or stable disease receive consolidation therapy comprising alemtuzumab subcutaneously on days 1-3. Treatment repeats weekly for up to 6 courses in the absence of disease progression.

Patients are followed at 2 months, every 3 months for 1 year, and then every 6 months for 7 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Specific Diagnosis of B-Cell CLL
* An absolute lymphocytosis of > 5,000/μL
* Morphologically, the lymphocytes must appear mature with < 55% prolymphocytes
* Bone marrow examination must include at least a unilateral aspirate and biopsy; the aspirate smear must show > 30% of all nucleated cells to be lymphoid or the bone marrow core biopsy must show lymphoid infiltrates compatible with marrow involvement by CLL; the overall cellularity must be normocellular or hypercellular
* Local institution lymphocyte phenotype must reveal a predominant B-cell monoclonal population sharing a B-cell marker (CD19, CD20, CD23) with the CD5 antigen, in the absence of other pan-T-cell markers; additionally, the B-cells must be monoclonal with regard to expression of either κ or λ and have surface immunoglobulin expression of low density; patients with bright surface immunoglobulin levels must have CD23 co-expression
* Patients must be in the intermediate- or high-risk categories of the modified three-stage Rai staging system (i.e., stages I, II, III, or IV)
* Patients in the intermediate-risk group must have evidence of active disease as demonstrated by at least one of the following criteria:

  * Massive or progressive splenomegaly, hepatomegaly and/or lymphadenopathy;
  * Presence of weight loss > 10% over the preceding 6 month period;
  * Grade 2 or 3 fatigue;
  * Fevers > 100.5°F or night sweats for greater than 2 weeks without evidence of infection;
  * Progressive lymphocytosis with an increase of > 50% over a 2 month period or an anticipated doubling time of less than 6 months
* No prior therapy for CLL including corticosteroids for autoimmune complications that have developed since the initial diagnosis of CLL
* No medical condition requiring chronic use of oral corticosteroids
* Performance Status 0 - 2
* Due to alterations in host immunity, patients with HIV may not be enrolled
* Due to the unknown teratogenic potential of alemtuzumab, pregnant or nursing women may not be enrolled; women and men of reproductive potential should agree to use an effective means of birth control
* Creatinine =< 1.5 x upper limit of institutional normal value
* Coomb's Testing NEGATIVE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2004-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lin, Principal Investigator — Cancer and Leukemia Group B
Locations (2):
- United States (2):
  - Cancer and Leukemia Group B, Chicago, Illinois
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- [Derived] Jones JA, Ruppert AS, Zhao W, Lin TS, Rai K, Peterson B, Larson RA, Marcucci G, Heerema NA, Byrd JC. Patients with chronic lymphocytic leukemia with high-risk genomic features have inferior outcome on successive Cancer and Leukemia Group B trials with alemtuzumab consolidation: subgroup analysis from CALGB 19901 and CALGB 10101. Leuk Lymphoma. 2013 Dec;54(12):2654-9. doi: 10.3109/10428194.2013.788179. Epub 2013 May 9. PMID 23547837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2005 and December 2006, 103 participants were recruited.
Pre-assignment Details: One participant was deemed ineligible and is excluded from all analyses per study design.
Groups:
- Alemtuzumab Consolidation: Alemtuzumab consolidation following fludarabine and rituximab induction in patients with B-cell CLL
Period: Overall Study
Arm/Group | Alemtuzumab Consolidation
Started | 102
Completed | 102
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab Consolidation
Number analyzed (Participants) | 102
Age, Continuous [Median (Full Range); unit: years] | 61 [23 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 75
Region of Enrollment [Number; unit: participants]
  United States | 102
Rai Stage [Number; unit: participants] — Rai staging is a way to categorize the disease progression of chronic lymphocytic leukemia (CLL); higher stages reflect increasing severity. Rai Stage 0: Lymphocytosis only, Rai Stage I: Lymphocytosis and lymphadenopathy, Rai Stage II: Lymphocytosis and hepatomegaly +/- splenomegaly, Rai Stage III: Lymphocytosis and anemia, Rai Stage IV: Lymphocytosis and thrombocytopenia
  participants
    Stage 0 | 1
    Stage I-II | 71
    Stage III-IV | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Complete Response After Treatment With Fludarabine & Rituximab Followed by Alemtuzumab
Description: A complete response, as defined by the National Cancer Institute Working Group (NCIWG):
  - CR: no lymphadenopathy, hepatomegaly, splenomegaly or constitutional symptoms; normal complete blood count; confirmed by bone marrow (BM) aspirate & biopsy
Time Frame: Duration of treatment (up to 13.5 months)
Population: 58 participants were treated with Alemtuzumab.
Measure: Number; unit: participants
Arm/Group | Alemtuzumab Consolidation
Number analyzed (Participants) | 58
participants | 38

2. Secondary Outcome: Number of Participants With a Complete or Partial Response After Induction Therapy With Fludarabine & Rituximab
Description: Response, as defined by the National Cancer Institute Working Group (NCIWG):
  CR: no lymphadenopathy, hepatomegaly, splenomegaly or constitutional symptoms; normal complete blood count; confirmed by bone marrow (BM) aspirate & biopsy
  PR: 50% decrease in peripheral blood lymphocytes, lymphadenopathy, liver/spleen size, presence/absence of constitutional symptoms; plus ≥1 of the following: ≥1500/μL polymorphonuclear leukocytes, >100,000/μL platelets, >11.0 g/dL hemoglobin or 50% improvement for these parameters without transfusions
Time Frame: Up to 9 months
Measure: Number; unit: participants
Arm/Group | Alemtuzumab Consolidation
Number analyzed (Participants) | 102
participants | 92

3. Secondary Outcome: 2 Year Progression Free Survival
Description: Percentage of patients who were alive and progression free at 2 years. The 2-year progression free survival was estimated using the Kaplan Meier method.
Time Frame: 2 years from registration
Measure: Number; unit: percentage of participants
Arm/Group | Alemtuzumab Consolidation
Number analyzed (Participants) | 102
percentage of participants | 72

4. Secondary Outcome: 2 Year Survival
Description: Percentage of participants who were alive at 2 years. The 2 year survival was estimated using the Kaplan Meier method.
Time Frame: 2 years from registration
Measure: Number; unit: percentage of participants
Arm/Group | Alemtuzumab Consolidation
Number analyzed (Participants) | 102
percentage of participants | 86

5. Secondary Outcome: Number of Participants With Severe Non-Hematologic Adverse Events During Treatment With Alemtuzumab
Description: The National Cancer Institute (NCI) Common Toxicity Criteria (CTC) Version 2.0 was used to evaluate toxicity. Severe Adverse events are defined as grade 3, 4 or 5, at least possibly related to treatment.
  Grade 1: mild; Grade 2: moderate; Grade 3: Severe; Grade 4: Life Threatening; Grade 5: Death.
Time Frame: 6 weeks beginning at study week 36
Population: 58 participants were treatment with Alemtuzumab.
Measure: Number; unit: participants
Arm/Group | Alemtuzumab Consolidation
Number analyzed (Participants) | 58
participants | 23

ADVERSE EVENTS:
Groups:
- FR Induction: Fludarabine and rituximab induction in pts with B-cell CLL
- Alemtuzumab Consolidation: Alemtuzumab consolidation following fludarabine and rituximab induction
Arm/Group | FR Induction | Alemtuzumab Consolidation
Serious Adverse Events (participants affected / at risk) | 19/102 | 23/58
Other Adverse Events (participants affected / at risk) | 101/102 | 55/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FR Induction (N=102) | Alemtuzumab Consolidation (N=58)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (6) | 7 (7)
Hemoglobin decreased (Blood and lymphatic system disorders) | 12 (13) | 20 (26)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Lymphatic disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (3)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (2)
Left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 4 (5)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (3)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7) | 7 (8)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4)
Chest pain (General disorders) | 2 (2) | 2 (2)
Chills (General disorders) | 4 (4) | 4 (4)
Edema limbs (General disorders) | 4 (4) | 3 (3)
Fatigue (General disorders) | 12 (12) | 19 (23)
Fever (General disorders) | 5 (5) | 9 (10)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 3 (3) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Visceral edema (General disorders) | 0 (0) | 1 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 3 (3)
Encephalomyelitis infection (Infections and infestations) | 1 (1) | 1 (1)
Infectious meningitis (Infections and infestations) | 0 (0) | 2 (2)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Opportunistic infection (Infections and infestations) | 0 (0) | 3 (4)
Pneumonia (Infections and infestations) | 2 (2) | 5 (7)
Sepsis (Infections and infestations) | 1 (1) | 8 (8)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 9 (11)
Alkaline phosphatase increased (Investigations) | 0 (0) | 6 (7)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 9 (11)
Blood bilirubin increased (Investigations) | 2 (2) | 5 (6)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1)
Creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 3 (4) | 5 (8)
Haptoglobin decreased (Investigations) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 3 (3) | 7 (9)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 5 (8)
Neutrophil count decreased (Investigations) | 13 (14) | 14 (20)
Platelet count decreased (Investigations) | 13 (14) | 18 (25)
Weight gain (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 5 (6)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 5 (6) | 11 (14)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Serum calcium decreased (Metabolism and nutrition disorders) | 3 (3) | 10 (12)
Serum glucose decreased (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Serum phosphate decreased (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2) | 10 (11)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 7 (8)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Mini mental status examination abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 4 (4)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (3)
Renal hemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 2 (2)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 10 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 6 (6) | 8 (9)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hematoma (Vascular disorders) | 0 (0) | 2 (2)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 6 (9)
Thrombosis (Vascular disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FR Induction (N=102) | Alemtuzumab Consolidation (N=58)
Blood disorder (Blood and lymphatic system disorders) | 1 (9) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (13) | 5 (6)
Hemoglobin decreased (Blood and lymphatic system disorders) | 73 (183) | 38 (89)
Hemolysis (Blood and lymphatic system disorders) | 2 (5) | 2 (2)
Lymph node pain (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (2) | 3 (6)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 1 (4)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 2 (5) | 1 (1)
Dry eye syndrome (Eye disorders) | 1 (1) | 1 (1)
Eye disorder (Eye disorders) | 4 (4) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Optic nerve edema (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 1 (2)
Vision blurred (Eye disorders) | 3 (3) | 1 (1)
Watering eyes (Eye disorders) | 4 (5) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (6) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 11 (18) | 3 (4)
Ascites (Gastrointestinal disorders) | 1 (3) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 29 (51) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 25 (34) | 18 (29)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (6) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 3 (5) | 4 (5)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 4 (6) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 4 (4) | 1 (2)
Nausea (Gastrointestinal disorders) | 58 (104) | 20 (24)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 24 (30) | 7 (7)
Chest pain (General disorders) | 8 (11) | 2 (4)
Chills (General disorders) | 28 (32) | 13 (15)
Edema limbs (General disorders) | 6 (9) | 6 (6)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 84 (200) | 44 (106)
Fever (General disorders) | 26 (33) | 14 (18)
Flu-like symptoms (General disorders) | 3 (4) | 0 (0)
Gait abnormal (General disorders) | 1 (1) | 0 (0)
General symptom (General disorders) | 1 (1) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 7 (7)
Localized edema (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 11 (11) | 6 (10)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 9 (9) | 4 (5)
Immune system disorder (Immune system disorders) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 2 (3) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4) | 5 (5)
Catheter related infection (Infections and infestations) | 0 (0) | 2 (3)
Conjunctivitis infective (Infections and infestations) | 2 (2) | 2 (2)
Cranial nerve infection (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 2 (2) | 1 (1)
Gallbladder infection (Infections and infestations) | 1 (1) | 0 (0)
Gastric infection (Infections and infestations) | 1 (1) | 0 (0)
Gingival infection (Infections and infestations) | 1 (1) | 1 (1)
Hepatic infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 4 (7) | 8 (11)
Infectious colitis (Infections and infestations) | 2 (2) | 1 (1)
Lip infection (Infections and infestations) | 3 (5) | 0 (0)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0)
Opportunistic infection (Infections and infestations) | 1 (1) | 2 (2)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (2) | 1 (1)
Pancreas infection (Infections and infestations) | 1 (1) | 0 (0)
Paranasal sinus infection (Infections and infestations) | 1 (1) | 0 (0)
Penile infection (Infections and infestations) | 0 (0) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 4 (5) | 0 (0)
Pneumonia (Infections and infestations) | 7 (11) | 5 (6)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1)
Scrotal infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 10 (11)
Sinusitis (Infections and infestations) | 10 (15) | 5 (8)
Skin infection (Infections and infestations) | 4 (5) | 2 (2)
Soft tissue infection (Infections and infestations) | 1 (1) | 3 (3)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 14 (18) | 11 (15)
Ureteritis (Infections and infestations) | 3 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (7) | 2 (3)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Biliary anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Small intestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Venous injury - Extremity-upper (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 18 (41) | 9 (19)
Alkaline phosphatase increased (Investigations) | 9 (11) | 8 (13)
Aspartate aminotransferase increased (Investigations) | 28 (60) | 10 (19)
Blood bilirubin increased (Investigations) | 16 (37) | 7 (16)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1)
Creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 20 (41) | 10 (23)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Haptoglobin decreased (Investigations) | 1 (1) | 0 (0)
Laboratory test abnormal (Investigations) | 9 (11) | 4 (6)
Leukocyte count decreased (Investigations) | 41 (97) | 22 (37)
Lymphocyte count decreased (Investigations) | 26 (68) | 15 (32)
Neutrophil count decreased (Investigations) | 78 (215) | 39 (96)
Platelet count decreased (Investigations) | 69 (194) | 33 (113)
Serum cholesterol increased (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 2 (5) | 0 (0)
Weight loss (Investigations) | 3 (3) | 3 (3)
Alkalosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 14 (15) | 8 (8)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 43 (118) | 18 (51)
Blood uric acid increased (Metabolism and nutrition disorders) | 6 (8) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 5 (6) | 1 (2)
Glucose intolerance (Metabolism and nutrition disorders) | 2 (7) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 6 (8) | 4 (4)
Serum calcium decreased (Metabolism and nutrition disorders) | 21 (34) | 13 (17)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 8 (8) | 3 (7)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 8 (9) | 4 (4)
Serum potassium decreased (Metabolism and nutrition disorders) | 9 (20) | 6 (6)
Serum potassium increased (Metabolism and nutrition disorders) | 7 (9) | 4 (4)
Serum sodium decreased (Metabolism and nutrition disorders) | 12 (18) | 7 (8)
Serum sodium increased (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Serum triglycerides increased (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (34) | 8 (12)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (25) | 5 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Joint disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (24) | 10 (12)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (20) | 3 (4)
Upper extremity dysfunction (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Tumor flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 11 (16) | 4 (5)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 27 (47) | 15 (19)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 2 (6)
Neurological disorder NOS (Nervous system disorders) | 3 (3) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 5 (5) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (16) | 3 (3)
Sinus pain (Nervous system disorders) | 1 (2) | 1 (2)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (2) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 7 (10) | 4 (7)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 13 (16) | 7 (10)
Insomnia (Psychiatric disorders) | 17 (26) | 9 (10)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder hemorrhage (Renal and urinary disorders) | 1 (1) | 2 (2)
Bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (painful urination) (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Renal and urinary disorders) | 5 (7) | 0 (0)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 6 (8) | 4 (4)
Urinary retention (Renal and urinary disorders) | 3 (4) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (3) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 7 (9)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (44) | 29 (43)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 (31) | 16 (27)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 6 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (6) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (8) | 3 (4)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (19) | 14 (20)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 48 (69) | 33 (57)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (5)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 21 (29) | 13 (22)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
Flushing (Vascular disorders) | 2 (2) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 1 (1)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 4 (7) | 3 (6)
Hypertension (Vascular disorders) | 6 (11) | 4 (8)
Hypotension (Vascular disorders) | 17 (24) | 6 (6)
Phlebitis (Vascular disorders) | 1 (2) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less